CLINICAL TRIAL: NCT05972226
Title: Self-care, Remote Monitoring and Elearning for Children and Young People With Asthma
Acronym: ASTHMAME
Status: Completed | Type: Observational
Sponsor: Sheffield Children's NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: SCH-2238
Record Dates: First submitted 2019-12-31; First posted 2023-08-02 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2019-12

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Asthma is a long-term condition in children, often managed by general practitioners (GPs) in primary care but some children with asthma need hospital treatment and care by experienced paediatricians and nurses. The positive effects of treatment for childhood asthma are well-documented however, less than 50% children take their medications regularly as prescribed. As well as causing poor control of asthma symptoms, failing to take medication as prescribed is a problem that is causing huge cost and wastage to the NHS.

Some of the barriers to taking medications as prescribed include people's beliefs about their illness or medications and forgetting or being too busy. These barriers can be addressed by providing education, reminders and incentives.

Monitoring medication usage is complex but studies have shown that use of electronic monitoring devices with education does improve the number of asthma attacks. Digital solutions for asthma self-care, including "smart-inhalers" that monitor medication usage and Apps for remote monitoring and self-management are likely to transform health services by providing supported self-management, prioritisation of the more unwell patients and reductions in hospital visits.

Asthma + me, a digital self-care solution has been developed by Aseptika Ltd, in consultation with Sheffield Children's Hospital, to support children with asthma. It uses a monitoring device that connects wirelessly to the Asthma +me App and monitors medication usage, providing education tips, reminders and incentives.

In this project, 15 children (and their families) will trial Asthma + me with a PUFFClicker and a 3-4 hour education session and report what worked and what didn't using structured interviews and questionnaires. At the same time the investigators will map out the number of patients that could potentially use this solution to self-manage their asthma, with the support of the hospital, until they are ready to be discharged back to their GP.

DETAILED DESCRIPTION:
Asthma is a long-term condition in children, often managed in primary care but around 20% children with asthma require secondary or tertiary level treatment and care by experienced respiratory paediatricians and nurses. The positive effects of treatment with inhaler and anti-inflammatory medications for childhood asthma are well-documented however, less than 50% children take their medications regularly as prescribed. Asthma deaths in children are rare but the national review of asthma deaths in the UK between 2012 and 2013 concluded that two thirds of the asthma deaths were preventable and that poor adherence to therapy was found to be a preventable cause in 34%.

It is known that educational interventions and use of written action plans improve asthma control. However, two thirds of patients do not attend their asthma review. Lack of adherence to medications is a global problem with £300million worth of medications /yr wasted in primary care due to poor adherence and 50% patients not taking medication as prescribed. With the UK facing an increasingly unmanageable demand on healthcare services, this morbidity and cost needs to be addressed.

So, why do people with asthma omit their medications? Clinicians have developed a conceptual framework to enable clinicians to understand the barriers to medication adherence. Habit formation is underpinned by a complex interaction of feedback, problem solving, prompts and implementation plans. The interaction between motivation (reasons that people "won't" take medication, such as illness perceptions, medication beliefs and contrivance) and capability opportunity (reasons that people "can't" take medication, such as forgetting, being too busy, having trouble incorporating into the routine) needs to be understood and addressed in order to change and sustain habit formation.

Adherence monitoring methods have been studied at length in patients with asthma, ranging from non-judgemental questioning by a clinician, which is cheap and easy to do in clinic, but vastly overestimates adherence, to self-report questionnaires and diary cards to prescription refill data and drug assays. These methods are increasingly objective, but remain subject to inaccuracies due to susceptibility to dose "dumping" and impracticalities. The most objective method of adherence monitoring is the use of electronic monitoring devices (EMDs) which can provide continuous monitoring and "smart" features such as transmission of data to electronic devices. The "STAAR" (Study of Asthma Adherence Reminders) study used adherence monitoring with feedback to target both motivation and capability opportunity with an educational/behavioural intervention and a practical adherence facilitator with reminder alarms chosen from a range of alarms by the child. Although a significant improvement in adherence from 49% to 70% was noted in the intervention group, there was no significant improvement in ACQ, the primary outcome measure. There was, however, a significantly lower number of exacerbations in the intervention group, measured by number of hospital and GP visits, number of courses of oral steroids and number of days missed from school.

There is a growing number of digital solutions for asthma Self-Care, with many of these produced by pharmaceutical companies as companion products or research tools. In addition, an increasing number of HealthApps and remote monitoring self-management software platforms are appearing on the commercial market. There are challenges to overcome before these can be implemented in paediatric clinical practice as all are adult based, are of variable quality, and more research is needed to refine the technology and links to electronic health records. However, smart inhalers and HealthApps in a digitally evolving NHS have the potential to support self-management of long-term conditions such as asthma at scale, to support digital transformation of health services to risk stratify according to need and to provide a personalised approach to care, thereby reducing emergency admissions and improving patient safety and quality of life.

Asthma + me, will be a comprehensive CE-marked technology-enabled self-care solution for children and young people with asthma and their parents has been developed by Aseptika Ltd, in consultation with Sheffield Children's Hospital, to support children with asthma to implement a new intermediate care pathway bridging the transition from hospital outpatient services back to primary care. It is specifically designed to meet the needs of children aged 5-18yrs and has two versions within the same App; a child-friendly view and a parent/carer view making it different from the many adult asthma management Apps available. It also supports integrated devices, medication diaries, trigger alerts and symptom scores. Core to Asthma +me is education, engagement and empowerment for children /young people and their parents. It has an in-built syllabus supported with an intensive half-day family training session to upskill those newly diagnosed.

Asthma + me supports a universal metered-dose inhaler tracker that connects wirelessly to the Asthma +me App counting inhaler doses, providing reminders to take the next dose and acting as an activity tracker for children too young or unable to wear an activity tracker at school. Patient-generated data will be used to incentivise adherence through a novel motivating rewards system.

A PDF report will be sent automatically from Asthma +me to the electronic patient record at Sheffield Children's Hospital. The consultant paediatrician or asthma nurse can remotely review progress or can access the patient-generated data in the event of an emergency consultation. Uniquely, as the child or their parent enters their data, their asthma action plan is automatically populated, viewed on the smart phone, printed and emailed as an integral part of the weekly report.

In this project, 15 children (and their families) will trial Asthma + me with PUFFClicker and 4 hour education session and report what worked and what didn't. The investigators will assess their views using structured Interviews and questionnaires and the investigators will look at any changes in their asthma symptoms. The investigators will also map patient pathways and collect health economics data to project costs and the number of patients that could potentially use this solution to self-manage their asthma, with the support of the hospital, until they are ready to be discharged back to their GP.

ELIGIBILITY:
Inclusion Criteria:

1. Age 5 to 15 years 11 months
2. Doctor-diagnosed asthma
3. Prescribed MDI inhalers
4. Asthma severity BTS level 3 or below.

Exclusion Criteria:

1. Non-English speaking families
2. Prescribed dry powder inhaler devices
3. Admission with acute asthma in the last 3 months

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Inclusion Criteria:
  1. Age 5 to 15 years 11 months
  2. Doctor-diagnosed asthma
  3. Prescribed MDI inhalers
  4. Asthma severity BTS level 3 or below.
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2018-07-16 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Acceptability | 17 months
  Acceptability of the Asthma and Me software, the PUFFClicker and the Education package, as assessed by the patient/parent, clinician and teacher using investigator designed questionnaires
Barriers to implementation of the Asthma and Me software | 17 months
  Barriers to implementation of the Asthma and Me software, the PUFFClicker and the Education package, as assessed by the patient/parent, clinician and teacher using investigator designed questionnaires

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Facility, Sheffield Childrens Hospital, Sheffield, United Kingdom